CLINICAL TRIAL: NCT03242759
Title: Non-Interventional Study (NIS) Collecting Experiences For IPF in Taiwan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0303
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with idiopathic pulmonary fibrosis (IPF)
  Interventions: Drug: nintedanib; Drug: pirfenidone

INTERVENTIONS:
Drug: nintedanib — Drug
  Other Names: OVEF
Drug: pirfenidone — Drug

SUMMARY:
This is a non-interventional, multi-center study to collect data from patients with idiopathic pulmonary fibrosis (IPF) in clinical practice in Taiwan. The study will be carried out at 10 medical centers, the expert centers where IPF patients are mainly managed in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients can be included if ALL the following criteria are met:

  1.Newly diagnosed with IPF within 6 months based upon recent ATS/ERS/JRS/ALAT IPF guideline (Ref 1, Raghu G, et al. 2011).
* Exclusion of other known causes of ILD (e.g. domestic and occupational environmental exposures, connective tissue disease, and drug toxicity).
* Assessment of IPF based on HRCT or HRCT and surgical lung biopsy, if available. 2.Patient ≥ 20 years of age 3.Written informed consent prior to participation 4.Patients with further follow-up possible with participating physician during planned study period 5.Ability to read and write in the local language

Exclusion Criteria:

* Patients should not be included if ANY of the following criteria is met:

  1. Lung transplantation expected within next 6 months.
  2. Inclusion in ongoing clinical trials.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out at 10 medical centers, the expert centers where idiopathic pulmonary fibrosis (IPF) patients are mainly managed in Taiwan.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional multi-center study based on newly collected data on idiopathic pulmonary fibrosis (IPF) patients in clinical practice in Taiwan with a planned 2-year followed-up period to characterize the IPF population in Taiwan with regard to their clinical course under clinical practice conditions in Taiwan.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug: Eligible patients with idiopathic pulmonary fibrosis (IPF) who signed the informed consent and fulfilled all inclusion criteria and no exclusion criteria, recruiting from 10 hospitals in Taiwan, and used anti-fibrotic drug were included in this group.
- Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug: Eligible patients with idiopathic pulmonary fibrosis (IPF) who signed the informed consent and fulfilled all inclusion criteria and no exclusion criteria, recruiting from 10 hospitals in Taiwan, and did not use anti-fibrotic drug were included in this group.
Period: Overall Study
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Started | 88 | 13
Completed | 53 | 6
Not Completed | 35 | 7
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Administrative problems | 1 | 1
Not completed — Death | 22 | 0
Not completed — Change visit schedule | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients: all patients who signed the informed consent and fulfilled all inclusion criteria and no exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug | Total
Number analyzed (Participants) | 88 | 13 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.7 (8.97) | 74.1 (10.64) | 74.6 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 0 | 17
  Male | 71 | 13 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Oriental | 88 | 13 | 101
Percent predicted Forced Vital Capacity (FVC) of lung function [Mean (Standard Deviation); unit: Percentage of predicted FVC] — Baseline measures of percentages of predicted Forced Vital Capacity of lung function (FVC) were shown.
  Percentage of predicted FVC | 69.7 (14.06) | 97.8 (10.97) | 73.3 (16.64)
Percent predicted Diffusing capacity of the Lungs for Carbon monoxide (DLco) of lung function [Mean (Standard Deviation); unit: Percentage of perdicted DLco] — Baseline measures of the percentages of predicted diffusing capacity of the Lungs for Carbon monoxide (DLco) were shown.
  Percentage of perdicted DLco | 42.7 (19.74) | 57.5 (17.96) | 45.2 (20.11)
Percent predicted oxygen saturation (SpO2) [Mean (Standard Deviation); unit: Percentage of predicted SpO2] — Baseline measures of percentages of predicted oxygen saturation (SpO2) were shown.
  Percentage of predicted SpO2 | 95.5 (2.31) | 97.5 (1.69) | 95.8 (2.33)
Percent predicted Total Lung Capacity (TLC) [Mean (Standard Deviation); unit: Percentage of perdicted TLC] — Baseline measures of the percentages of predicted Total Lung Capacity (TLC) were shown.
  Percentage of perdicted TLC | 74.3 (13.25) | 100.2 (13.04) | 77.2 (15.50)
Percent predicted Inspiratory Capacity (IC) [Mean (Standard Deviation); unit: Percentage of perdicted IC] — Baseline measures of the percentages of predicted Inspiratory Capacity (IC) were shown.
  Percentage of perdicted IC | 62.8 (15.62) | 87.5 (21.49) | 65.6 (17.87)

OUTCOME MEASURES:

1. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Forced Vital Capacity (FVC) at Week 52
Description: Annual Change from Baseline in percentage of predicted Forced Vital Capacity (FVC) at Week 52 was reported.
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted FVC
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted FVC | -0.5 (10.78) | 4.1 (7.73)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.505, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.181, Paired t-test

2. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Forced Vital Capacity (FVC) at Week 100
Description: Annual Change from Baseline in percentage of predicted Forced Vital Capacity (FVC) at Week 100 was reported.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted FVC
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted FVC | -0.2 (7.74) | -2.5 (4.52)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.571, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.232, Paired t-test

3. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Diffusing Capacity of the Lungs for Carbon Monoxide (DLco) at Week 52
Description: Annual Change from Baseline in percentage of predicted Diffusing capacity of the Lungs for Carbon monoxide (DLco) at Week 52 was reported
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted DLco
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted DLco | -7.3 (10.47) | -2.8 (8.27)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.375, Paired t-test

4. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Diffusing Capacity of the Lungs for Carbon Monoxide (DLco) at Week 100
Description: Annual Change from Baseline in percentage of predicted Diffusing capacity of the Lungs for Carbon monoxide (DLco) at Week 100 was reported.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted DLco
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted DLco | 0.5 (6.83) | -2.6 (6.26)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.027, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.938, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Oxygen Saturation (SpO2) at Week 52
Description: Annual Change from Baseline in percentage of predicted oxygen saturation (SpO2) at Week 52 was reported.
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted SpO2
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted SpO2 | -0.8 (2.22) | -0.8 (0.92)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.048, Paired t-test

6. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Oxygen Saturation (SpO2) at Week 100
Description: Annual Change from Baseline in percentage of predicted oxygen saturation (SpO2) at Week 100 was reported.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted SpO2
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted SpO2 | -0.2 (0.96) | -0.6 (0.84)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.018, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.125, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Total Lung Capacity (TLC) at Week 52
Description: Annual Change from Baseline in percentage of predicted Total Lung Capacity (TLC) at Week 52was reported.
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted TLC
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted TLC | -0.4 (9.97) | -1.4 (12.18)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.073, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.755, Paired t-test

8. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Total Lung Capacity (TLC) at Week 100
Description: Annual Change from Baseline in percentage of predicted Total Lung Capacity (TLC) at Week 100 was reported.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted TLC
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted TLC | -2.3 (3.76) | -3.4 (6.89)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.281, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Inspiratory Capacity (IC) at Week 52
Description: Annual Change from Baseline in percentage of predicted Inspiratory Capacity (IC) at Week 52 was reported.
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted IC
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted IC | -6.8 (10.18) | -6.1 (1.73)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.008, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Annual Change From Baseline in Percentage of Predicted Inspiratory Capacity (IC) at Week 100
Description: Annual Change from Baseline in percentage of predicted Inspiratory Capacity (IC) at Week 100 was reported.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage of predicted IC
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Percentage of predicted IC | -4.5 (5.00) | -6.0 (2.40)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.031, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Time to First Acute Exacerbation of Idiopathic Pulmonary Fibrosis
Description: Time to first acute exacerbation of idiopathic pulmonary fibrosis was reported.
Time Frame: From baseline until end of follow-up, up to 899 days.
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Days | 497.0 [6.0 to 751.0] | 521.5 [111.0 to 721.0]

12. Secondary Outcome: Annual Change in Total Score of St. Georges Respiratory Questionnaire (SGRQ) at Week 52
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. The questionnaire included 3 subscales measures: symptoms, activity limitation, and social, and emotional impact of disease (each subscale score ranges from 0 to 100 with higher score indicating poorer quality of life). The SGRQ total score was calculated by summing weights from all positive items, divided by sum of weights for all items in SGRQ questionnaire and multiplying by 100. The total score of SGRQ ranged from 0 (no effect on quality of life) to 100 (maximum perceived distress). Thus, a higher score indicated a poorer quality of life. Annual change in score of St. Georges Respiratory Questionnaire (SGRQ) at Week 52 was reported.
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Score on a scale | 8.4 (16.52) | 0.2 (8.12)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p < 0.001, Paired t-test
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.939, Paired t-test

13. Secondary Outcome: Annual Change in Total Score of St. Georges Respiratory Questionnaire (SGRQ) at Week 100
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. The questionnaire included 3 subscales measures: symptoms, activity limitation, and social, and emotional impact of disease (each subscale score ranges from 0 to 100 with higher score indicating poorer quality of life). The SGRQ total score was calculated by summing weights from all positive items, divided by sum of weights for all items in SGRQ questionnaire and multiplying by 100. The total score of SGRQ ranged from 0 (no effect on quality of life) to 100 (maximum perceived distress). Thus, a higher score indicated a poorer quality of life. Annual change in score of St. Georges Respiratory Questionnaire (SGRQ) at Week 100 was reported.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Score on a scale | 2.6 (13.36) | 1.6 (6.17)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.169, Paired t-test
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.545, Paired t-test

14. Secondary Outcome: Annual Change in Score of Chronic Obstructive Pulmonary Disease Assessment Test (CAT) at Week 52
Description: The Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) is an 8-item, health status instrument which provides a method for assessing the impact of COPD on the patient's health and quality of life. The CAT score (ranging from 0 to 40) was calculated for each individual by summing the points for each item. A decrease in CAT score represents an improvement in health status, whereas an increase in CAT score represents a worsening in health status.
Time Frame: At baseline and Week 52
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Score on a scale | 1.4 (7.80) | 0.2 (1.96)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.333, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.786, Paired t-test

15. Secondary Outcome: Annual Change in Score of Chronic Obstructive Pulmonary Disease Assessment Test (CAT) at Week 100
Description: as for outcome 14
Time Frame: At baseline and Week 100
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Score on a scale | 0.7 (4.37) | 0.7 (2.13)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.245, Paired t-test
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.454, Paired t-test

16. Secondary Outcome: Annual Change in Six-Minute Walk Test (6MWT) at Week 52
Description: Annual change in Six-Minute Walk Test (6MWT) at Week 52 was reported. The 6MWT measured the distance that a person can walk in 6 minutes, providing information regarding functional capacity, response to therapy and prognosis.
Time Frame: At baseline and Week 52.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Meter | -7.6 (60.42) | 7.1 (31.53)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.543, Paired t-test
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.733, Paired t-test

17. Secondary Outcome: Annual Change in Six-Minute Walk Test (6MWT) at Week 100
Description: Annual change in Six-Minute Walk Test (6MWT) at Week 100 was reported. The 6MWT measured the distance that a person can walk in 6 minutes, providing information regarding functional capacity, response to therapy and prognosis.
Time Frame: At baseline and Week 100.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Meter | -20.7 (36.60) | -2.3 (20.51)
Statistical Analysis 1: Comparison: Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.046, Paired t-test
Statistical Analysis 2: Comparison: Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug; Intra-group difference comparing to baseline was analyzed; Test type: Other; p = 0.898, Paired t-test

18. Secondary Outcome: Overall Survival
Description: Overall survival was reported. Overall survival was defined as the time from randomization to death due to any cause.
Time Frame: From baseline until end of follow-up, up to 899 days.
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 88 | 13
Days | 686.0 [14.0 to 899.0] | 641.0 [111.0 to 721.0]

19. Secondary Outcome: Number of Participants Per Death Reason Categories
Description: Number of participants per death reason categories was reported.
Time Frame: From baseline until end of follow-up, up to 899 days.
Population: All eligible patients who died during the study. All eligible patients: all patients who signed the informed consent and fulfilled all inclusion criteria and no exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
Number analyzed (Participants) | 28 | 1
Participants
  Related to idiopathic pulmonary fibrosis | 11 | 0
  Related to comorbidity | 7 | 1
  Other | 4 | 0
  Unknown | 6 | 0

ADVERSE EVENTS:
Time Frame: From baseline until end of follow-up, up to 899 days.
Description: All eligible patients: all patients who signed the informed consent and fulfilled all inclusion criteria and no exclusion criteria.
Arm/Group | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug
All-Cause Mortality (participants affected / at risk) | 28/88 | 1/13
Serious Adverse Events (participants affected / at risk) | 29/88 | 2/13
Other Adverse Events (participants affected / at risk) | 36/88 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug (N=88) | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug (N=13)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Death (General disorders) | 10 | 0
Pyrexia (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 0
Aspartate aminotransferase abnormal (Investigations) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idiopathic Pulmonary Fibrosis With Anti-fibrotic Drug (N=88) | Idiopathic Pulmonary Fibrosis Without Anti-fibrotic Drug (N=13)
Diarrhoea (Gastrointestinal disorders) | 29 | 0
Alanine aminotransferase abnormal (Investigations) | 10 | 1
Aspartate aminotransferase abnormal (Investigations) | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT03242759/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03242759/SAP_001.pdf